CLINICAL TRIAL: NCT00348517
Title: An Evaluation of the Safety and Efficacy of Systane Free FID 105783
Brief Title: Safety/Efficacy of Systane Free vs Refresh Liquigel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-05-45
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Systane (Experimental)
  Interventions: Other: Systane Free Lubricant Eye Drops
- Refresh (Active Comparator)
  Interventions: Other: Refresh Liquigel Lubricant Eye Drops

INTERVENTIONS:
Other: Systane Free Lubricant Eye Drops — 1-2 drops per eye four times per day for 42 days
  Arms: Systane
Other: Refresh Liquigel Lubricant Eye Drops — 1-2 drops per eye four times per day for 42 days
  Arms: Refresh

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of Systane Free FID 105783 when compared to Refresh Liquigel Lubricant Eye Drops (Allergan) in a specified population of dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

* >/= 3 corneal staining score using NEI scoring system.
* Need artificial tears at least some of the time.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* History or evidence of ocular or intraocular surgery in either eye within the past six months.
* History of intolerance or hypersensitivity to any component of the study medication.
* Use of Restasis within 30 days of Visit 1.
* Participation in an investigational drug or device study within 30 days of entering this study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11

PRIMARY OUTCOMES:
Change in corneal staining at Day 28 from baseline (Day 0) | Day 28